CLINICAL TRIAL: NCT05610579
Title: The 24 Hour Effects of Remedial Exercises With and Without Compression Therapy on Breast Cancer-related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Turkan Akbayrak, Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA22053
Record Dates: First submitted 2022-11-03; First posted 2022-11-09 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Lymphedema, Breast Cancer
Keywords: compression therapy; lymphedema; exercise
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema; Motor Activity | interventions — Exercise Therapy; Compression Bandages

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remedial exercises with compression bandage (Experimental)
  Interventions: Other: Remedial exercise; Other: Compression bandage
- remedial exercises (Active Comparator)
  Interventions: Other: Remedial exercise

INTERVENTIONS:
Other: Remedial exercise — Remedial exercise program will be taught by qualified physiotherapist. Patients will be practiced to the exercise 3 sets of 15 repetitions without compression. Patients will be monitored telephonically in the washout period for remain the routine activities.
Other: Compression bandage — Multi-layered short stretch bandaging will be applied for 23 hour. Patients will be practiced to the exercise 3 sets of 15 repetitions with compression bandage. The bandage will be removed at the same time the next day. Patients will be monitored telephonically in the washout period for remain the routine activities.
  Arms: remedial exercises with compression bandage

SUMMARY:
The aim of this study to investigate 24 hours of effects of remedial exercises with and without compression therapy on severity of lymphedema and symptoms of the lymphedema The present study is designed as a non-drug clinical trial. The patients will complete two remedial exercise sessions, one without and one with compression in a randomized order separated by a 3-day wash-out period.The main questions it aims to answer are

1. The 24 hour effects of remedial exercises with and without compression therapy on the severity of lymphedema are different in individuals with lymphedema associated with breast cancer surgery.
2. The 24 hour effects of remedial exercises with and without compression therapy on the symptoms of lymphedema are different in individuals with lymphedema associated with breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unilateral arm lymphedema related to breast cancer disease- Age between 18 and 75 years
* 2 cm or greater difference between the affected and unaffected arms in women with breast cancer related lymphedema
* At least 12 months after breast cancer surgery end

Exclusion Criteria:

* current recurrence of breast cancer
* bilateral involvement
* active infection
* presence of metastases
* diabetes mellitus
* hypertension
* pre-existing neuromusculoskeletal and neurological conditions
* edema due to other reasons (e.g., primary lymphedema, lung and heart diseases)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic measurements | Change in symptoms related to lymphedema from baseline up to end of 24 hour
  Ultrasound imaging was performed using a 5-13-Megahertz linear probe. During the procedure, the participants will be seated with their forearms supinated and extended on a pillow. Measurements will be made bilaterally from 10 cm distal and proximal to the elbow bend, from the midpoint of the medial and lateral epicondyles, along the line parallel to the arm axis.
Circumference measurement | Change in symptoms related to lymphedema from baseline up to end of 24 hour
  The severity of lymphedema between the two extremities will be measured by measuring the environment at 5 cm intervals.
Bioimpedance spectroscopy | Change in symptoms related to lymphedema from baseline up to end of 24 hour
  The patient is in the supine position with his arms and legs not touching each other. This measurement will be made using the Impedimed L-Dex U 400 device. The reference point is the top of both hands and the dorsum of the foot. This measurement is made using superficial electrodes and there is no risk. The percentage of fluid will be calculated by making a measurement for both arms.

SECONDARY OUTCOMES:
symptoms of lymphedema | Change in symptoms related to lymphedema from baseline up to end of 24 hour
  Four participant-reported lymphedema symptoms were assessed: swelling, heaviness, tightness commonly associated with BCRL. Using a 100 mm visual analogue scale (VAS), participants marked on it the extent to which they perceived their arm to be swollen, heavy or tight and pain during the past month, with 0 being "not at all" and 10 being "extremely".

CONTACTS AND LOCATIONS:
Locations (1):
- Gülbala Nakip, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McNeely ML, Campbell K, Ospina M, Rowe BH, Dabbs K, Klassen TP, Mackey J, Courneya K. Exercise interventions for upper-limb dysfunction due to breast cancer treatment. Cochrane Database Syst Rev. 2010 Jun 16;(6):CD005211. doi: 10.1002/14651858.CD005211.pub2. PMID 20556760
- [Result] McNeely ML, Campbell KL, Courneya KS, Mackey JR. Effect of acute exercise on upper-limb volume in breast cancer survivors: a pilot study. Physiother Can. 2009 Fall;61(4):244-51. doi: 10.3138/physio.61.4.244. Epub 2009 Nov 12. PMID 20808486
- [Result] Stout Gergich NL, Pfalzer LA, McGarvey C, Springer B, Gerber LH, Soballe P. Preoperative assessment enables the early diagnosis and successful treatment of lymphedema. Cancer. 2008 Jun 15;112(12):2809-19. doi: 10.1002/cncr.23494. PMID 18428212
- [Result] De Vrieze T, Vos L, Gebruers N, Tjalma WAA, Thomis S, Neven P, Nevelsteen I, De Groef A, Vandermeeren L, Belgrado JP, Devoogdt N. Protocol of a randomised controlled trial regarding the effectiveness of fluoroscopy-guided manual lymph drainage for the treatment of breast cancer-related lymphoedema (EFforT-BCRL trial). Eur J Obstet Gynecol Reprod Biol. 2018 Feb;221:177-188. doi: 10.1016/j.ejogrb.2017.12.023. Epub 2017 Dec 16. PMID 29277358
- [Result] Svensson BJ, Dylke ES, Ward LC, Black DA, Kilbreath SL. Screening for breast cancer-related lymphoedema: self-assessment of symptoms and signs. Support Care Cancer. 2020 Jul;28(7):3073-3080. doi: 10.1007/s00520-019-05083-7. Epub 2019 Oct 22. PMID 31641870
- [Result] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Result] Ricci V, Ricci C, Gervasoni F, Andreoli A, Ozcakar L. From histo-anatomy to sonography in lymphedema: EURO-MUSCULUS/USPRM approach. Eur J Phys Rehabil Med. 2022 Feb;58(1):108-117. doi: 10.23736/S1973-9087.21.06853-2. Epub 2021 Apr 16. PMID 33861039